CLINICAL TRIAL: NCT04647136
Title: The Effect of Fertility Health Awareness Strategies on Fertility Knowledge and Childbearing in Young Married Couples (FertStart)
Brief Title: The Effect of Fertility Health Awareness Strategies on Fertility Knowledge and Childbearing in Young Married Couples
Acronym: FertStart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: KK Women's and Children's Hospital (Other Government); Singapore Health Services (Other); Duke-NUS Graduate Medical School (Other); Cardiff University (Other); National Population and Talent Division (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 7.0
Record Dates: First submitted 2020-09-16; First posted 2020-11-30 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Fertility Awareness; Childbearing Intentions
Keywords: Fertility awareness; Attitudes; Intentions; Fertility screening; Couples
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fertility Health Screening (Active Comparator): Clinic-based fertility health screening and counselling
  Interventions: Diagnostic Test: Fertility Health Screening
- Fertility Awareness Tools (Active Comparator): Online intervention to provide fertility education and behavioural nudge for optimal reproductive timing.
  Interventions: Behavioral: Fertility Awareness Tools
- Control (No Intervention): No intervention

INTERVENTIONS:
Diagnostic Test: Fertility Health Screening — Basic fertility health screening comprising an anti-Mullerian hormone (AMH) test and semen analysis, a doctor's consultation to explain the results, and standardised reproductive counselling by a trained nurse comprising a discussion of reproductive plans (including addressing barriers the couple face), education on age-related fertility decline and limitations of artificial reproductive technologies, advice on the optimal reproductive timing and when to seek further help. An educational brochure will be handed to the couple during the counselling session.
  Arms: Fertility Health Screening
Behavioral: Fertility Awareness Tools — Online intervention consisting of 1) video targeting fertility education and specific attitudes, social norms and perceived control for having children, 2) a fertility awareness tool (FERTISTAT) and 3) an educational brochure on fertility. This intervention can be self-administered and is therefore easily scalable.
  Arms: Fertility Awareness Tools

SUMMARY:
Singapore, like many developed countries, is experiencing low birth rates, which is coupled with increasing age at first marriage and birth. In addition, demand for assisted reproduction technology treatments has increased over the years. Fertility awareness surveys have consistently shown that public awareness of age-related fertility decline and the limitations of fertility treatments is generally low, and this may lead to couples not optimising their fertility potential to achieve their family aspirations. This trial aims to study the effect of fertility health screening and fertility awareness tools on knowledge, attitudes and practice around childbearing among young Singaporean married couples.

ELIGIBILITY:
Inclusion Criteria:

* Married couple
* Both partners should be Singapore Citizens or Permanent Residents
* Female partner is 25 - 34 years old at time of recruitment
* Both partners agreeable and able to complete study procedures

Exclusion Criteria:

* Already have children, including from previous marriages
* Pregnant
* Currently undergoing or had previously went for any fertility evaluation and/or treatments
* Self-reported history of previous ectopic pregnancy in the female partner
* At least 1 partner unable to complete a self-administered questionnaire in English

Ages: 25 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 841 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Change in parenthood intentions | Baseline (before intervention) and 6 months later
  The difference in the female partner's intended age at first birth at 6 months post-randomization compared to baseline, elicited by a direct question in pre and post-questionnaires.

SECONDARY OUTCOMES:
Change in fertility awareness | Baseline (before intervention) and 6 months later
  The difference in fertility awareness as measured by the Cardiff Fertility Knowledge Scale (CFKS) at 6 months post-randomization compared to baseline. The CFKS is a 13-item scale where each correct answer is assigned 1 point. Points are summed and converted to the % correct fertility knowledge score with a range of 0 - 100%.
Conception efforts | 6 moths post-randomization
  Proportion of couples who are (a) attempting to conceive, (b) pregnant, (c) who pursued more comprehensive fertility screening and/or (d) who pursued fertility treatment.
Birth number | 2 and 3 years post-randomization
  Number of births
Birth timing | 2 and 3 years post-randomization
  Time to first birth

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan SL, Thumboo J, Boivin J, Saffari SE, Yin S, Yeo SR, Chan JKY, Ng KC, Chua KH, Yu SL. Effect of fertility health awareness strategies on fertility knowledge and childbearing in young married couples (FertStart): study protocol for an effectiveness-implementation hybrid type I multicentre three-arm parallel group open-label randomised clinical trial. BMJ Open. 2022 Jan 3;12(1):e051710. doi: 10.1136/bmjopen-2021-051710. PMID 34980614